CLINICAL TRIAL: NCT03277625
Title: Safety and Efficacy of Modified Single-loop Omega-shaped Reconstruction After Pancreaticoduodenectomy in Patients With High-risk Pancreas
Brief Title: Modified Reconstruction for Pancreatic Head Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Josef Hospital Bochum (Other)
Responsible Party: Principal Investigator, Orlin Belyaev, PD Dr. med., St. Josef Hospital Bochum
Other Study IDs: 16-5706
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Pancreaticoduodenal; Fistula
Keywords: pancreaticoduodenectomy
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pancreaticoduodenectomy: patients undergoing pancreticoduodenectomy and having a soft, fragile and/or fatty pancreatic remnant, combined with small pancreatic duct having a Diameter <3 mm.
  Interventions: Procedure: modified omega-shaped single-loop

INTERVENTIONS:
Procedure: modified omega-shaped single-loop — A double-layer, end-to-side, duct-to-mucosa PJ using interrupted polydioxanone 5-0 suture (PDS II, Ethicon, Somerville, USA) for the outer layer and interrupted polypropylene 5-0 suture (Prolene, Ethicon, USA) for the inner layer is the standard technique during PD at our Institution. For the modified omega-shaped single-Loop reconstruction the loop between PJ and HJ is left intentionally longer at about 25-30 cm and an additional side-to-side jejunojejunal anastomosis is performed at the lowest point between the afferent and efferent loops of the HJ This intestinal anastomosis is done in a double-layer continuous PDS 5-0 suture technique. Neither sealants, nor stents are being applied at the PJ. In cases of thin walled and tiny hepatic ducts, the HJ is splinted using an externally diverted T-tube.

SUMMARY:
This observational study aims to prove the safety and efficacy of a modified method of reconstruction after pancreatic head resection utilizing a single Omega shaped intestinal Loop with an additional anastomosis between the pancreatic and biliary anstomoses. This simple and fast method is expected to provide the advantages of a double-loop reconstruction without adding time and difficulty to the reconstruction process during pancreaticoduodenectomy. The additional intestinal anastomosis should allow Diversion of pancreatic Juice from bile thus reducing the severity of possible postoperative pancreatic Fistula, especially in the subgroup of patients undergoing a pancreaticoduodenectomy and having a high-risk pancreatic remnant, i.e. very soft, fragile and fatty pancreas with a tiny, non-dilated pancreatic main duct. The Primary Point of the study ist the severity of postoperative pancreatic Fistula, as well as the total rate of severe postoperative complications, defined as Grade 3b or more according to the classification of Dindo-Clavien.

DETAILED DESCRIPTION:
Postoperative pancreatic fistula (POPF) is the most common and specific complication of pancreaticoduodenectomy (PD) with reported rates of over 20% even at high-volume centers. POPF may cause life-threatening secondary complications such as postpancreatectomy hemorrhage (PPH), intraabdominal abscess, and sepsis, leading to increased costs, prolonged hospital stay as well as to delayed chemotherapy in oncologic patients.

A myriad of innovations in surgical technique has been introduced over the last several decades in order to reduce the rate and severity of POPF. One of these includes the double-loop (DL) reconstruction with isolated Roux-en-Y loops for the pancreatic and biliary anastomoses. It was first described in 1976 by Machado and has afterwards been applied by many surgeons in different variations. The method is based on the empirical hypothesis that diverting bile away from pancreatic juice may prevent their mutual activation and thus decrease their aggressiveness and detrimental effect on the pancreaticojejunostomy (PJ). Theoretically, reduction in the rate and severity of POPF should be expected. Some randomized controlled trials (RCT) reported decreased severity of POPF and lower rates of associated morbidity, whereas others failed to confirm these positive results. A substantially prolonged duration of surgery was observed in most of the studies.

In order to reduce the rate and severity of POPF without prolonging duration of surgery, we introduced in 2015 a new method of reconstruction during PD using a single long intestinal loop with a side-to-side anastomosis between the afferent and efferent limbs of the hepaticojejunostomy (HJ) similar to a Braun anastomosis in a Billroth II resection. It aimed at increasing the distance between the pancreatic and biliary anastomotic sites and facilitating isolated flow of bile and pancreatic secretions in a simple, fast and straightforward manner without the need for a time-consuming and sometimes technically challenging DL reconstruction.

This study aims to reveal how the new modified single-loop (mSL) method of reconstruction compares to the conventional single loop (SL) and DL methods in terms of severity and rate of POPF as well as associated major complications after PD in high-risk patients with a soft pancreatic remnant and a small pancreatic duct.

ELIGIBILITY:
Inclusion Criteria:

* pancreaticoduodenectomy
* soft, fragile or fatty pancreatic remnant combined with pancreatic duct <3mm

Exclusion Criteria:

* soft pancreas, but large pancreatic duct>3mm
* small pancreatic duct <3mm, but hard pancreatic remnant

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients undergoing elective and emergency pancreaticoduodenectomy irrespective of diagnosis. the typical Patient is an obese, old, has a small pancreatic lesion, either cystic or solid, not leading to obstruction of the pancreatic duct or the biliary duct.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Severity of postoperative pancreatic fistula | from postoperative day 3 until postoperative day 30
  grade B and grade C Fistula as clinically relevant

SECONDARY OUTCOMES:
Major postoperative complications | postoperative days 1 to 30
  all type of postoperative complications grades 3b, 4 and 5 (mortality) after Dindo-Clavien

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, St. Josef Hospital, Ruhr University of Bochum, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No